CLINICAL TRIAL: NCT00106821
Title: An 8 Week Randomized, Placebo Controlled, Double-blind Study to Assess the Efficacy of Tiotropium Inhalation Capsules in Patients of African Descent With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of Tiotropium in Patients of African Descent With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.294
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: Tiotropium Bromide Inhalation Powder

SUMMARY:
The purpose of this study is to look at the benefits of tiotropium, an approved drug for the treatment of bronchospasm associated with COPD (chronic obstructive pulmonary disease), in a population of patients with COPD who are of African American descent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of African descent
* 40 years of age or older
* Diagnosis of COPD
* History of smoking at least one pack per day for at least 10 years
* Currently experiencing shortness of breath at least with exertion

Exclusion Criteria:

* Asthma
* Recent myocardial infarction or hospitalization for congestive heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be FEV1 AUC (0-3) after 8 weeks of treatment

SECONDARY OUTCOMES:
FEV1 AUC0-3 after single dose, 4 weeks of treatment, peak FEV1 on each test day, trough FEV1 at weeks 4 & 8, FVC trough (weeks 4 & 8), peak and AUC(0-3) (on all test days), FEV1 and FVC at all time points, rescue albuterol use, dyspnea SOP questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (19):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Cooper Green Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - David Geffen School of Medicine, Los Angeles, California
  - VA Greater Los angeles Health Care Systems, Sepulveda, California
  - Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - Yale Univ. Pulmonary and Critical Care Medicine, West Haven, Connecticut
  - Emerald Coast Research Associates, Panama City, Florida
  - Bay Pines V. A. Medical Center, Saint Petersberg, Florida
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - LSU MC-Sheveport, Shreveport, Louisiana
  - Bronx VA Medical Center, The Bronx, New York
  - Brody School of Medicine, East Carolina University, Greenville, North Carolina
  - Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Attention: Amir Sharafkhaneh, M.D., Houston, Texas
  - VAMC Houston, Houston, Texas